CLINICAL TRIAL: NCT01308203
Title: Lipid Efficacy and Effects on HDL-C Metabolism of the Extended Release Niacin/Laropiprant Combination Added to Usual Therapy in Patients With Cardiovascular Disease and Low HDL-C That Did Not Achieve the Optional Very Low LDL-C Goal
Brief Title: Lipid Efficacy of the Extended Release Niacin/Laropiprant Combination in Patients With Cardiovascular Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Merck has decided to discontinue all studies with extended-release niacin/laropiprant.because the HPS2-THRIVE did not meet its primary endpoint
Sponsor: Daniel A. Siniawski (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Daniel A. Siniawski, Associated Medical Doctor, Hospital Italiano de Buenos Aires
Organization: Hospital Italiano de Buenos Aires (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1608
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Dyslipidemias
MeSH Terms: conditions — Coronary Artery Disease; Dyslipidemias | interventions — MK-0524

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended release niacin /laropiprant (Experimental): The patients will be randomized to one of two arms. The intervention is with the extended release niacin laropiprant combination, that is an add on of the usual medication that the primary care physician gave them to treat their lipid disorder (statin, ezetimibe or the combination of both).
  Interventions: Drug: Extended release niacin/laropiprant
- placebo (Placebo Comparator): The patients will received placebo added to the usual therapy their primary care physician gave them to treat their lipid disorder (statin, ezetimibe or the combination of both).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Extended release niacin/laropiprant — Randomized patient will received 1 tablet of 1g ERN/20 mg LRPT for the first 4 weeks of treatment. At week 4 (± 2 days)the patient will be assessed in the outpatient clinic. Patients with good tolerance to the study medication will receive 2 tablets of 1 g ERN/20 mg LRPT that should be taken together for the next 8 weeks. At week 12 (± 2 days), patients will be assessed in the outpatient clinic patients and will be crossed over to placebo.
  Arms: Extended release niacin /laropiprant
Drug: placebo — Randomized patient will received 1 oral 1 g tablet of placebo for the first 4 weeks of treatment. At week 4 (± 2 days), after randomization the patient will be assessed in the outpatient clinic. Patients with good tolerance to the study medication will receive 2 oral 1 g tablets of placebo that should be taken together for the next 8 weeks. At week 12 (± 2 days), patients will be assessed in the outpatient clinic patients and will be crossed over to active medication.
  Arms: placebo

SUMMARY:
* Clinical studies with statins have shown that patients that suffered a cardiovascular event have a high residual risk. Residual risk decreases with the attaining of progressive lower LDL-C levels.
* In patients treated with statins, HDL-C level is an independent inverse predictor of subsequent CV and coronary plaque progression, even when LDL-C levels are less than 70 mg/dL.
* Therefore the purpose on this study is to assess the lipid efficacy on lipid profile and effects on HDL-C metabolism and function of the extended release niacin/laropiprant combination added to usual therapy in very high risk patients with cardiovascular disease and low HDL-C that did not achieve the optional very low LDL-C or non-HDL-C goals

DETAILED DESCRIPTION:
During the screening period, patients will be pre-selected from medical records of patients that met the inclusion criteria. Patients who fulfilled the eligibility criteria will be invited to participate in the study by signing the consent form. After consenting, a screening blood sample test will be taken to determine TC, HDL-C, TG, LDL-C, non-HDL-C (the difference between TC and HDL-C), ALT, AST, CK, hemoglobin A1c (HbA1c), uric acid and TSH in the local laboratory. Patients who have HDL-C, LDL-C and/or non-HDL-C within inclusion criteria and had none of the biochemical exclusion criteria will be randomized one week after the screening blood test. Further blood samples will be obtained at baseline, 4 weeks (± 2 days), 12 weeks (± 2 days), 16 weeks (± 2 days) and 24 weeks (± 2 days). The blood samples will be centrifuged a 2000 rpm and a tube with blood serum will be sent to the local laboratory for measuring plasma levels of TC, HDL-C, TG, LDL-C, ALT, AST, CK, fasting glucose, HbA1c, creatinine, uric acid, ApoB, ApoA, Lp(a), high sensibility-C Reactive Protein (hs-CRP) and HDL-C sub-fractions (baseline, weeks 12 and 24). ALT, AST, CK, fasting glucose, creatinine and uric acid will be measured at weeks 4 and 16. A second tube will be frozen in -70ºC refrigerator an will be sent to the Department of Clinical Biochemistry of the Faculty of Pharmacy and Biochemistry from the University of Buenos Aires (Argentina) to determine: paraoxonase 1/arylesterase activity (PON1), soluble cell adhesion molecule level (ICAM-1), tumor necrosis factor-α (TNF-α), lipoprotein-associated phospholipase A2 (Lp-PLA2) and cholesterol ester transfer protein (CETP) activity. A third tube will be frozen in -70ºC refrigerator an will be sent to the Cardiovascular Research Center of the Faculty of Medical Sciences from the University of La Plata (Argentina) to determine ex vivo cellular cholesterol efflux capacity.

A unique patient number will be provided by the randomization coordinating centre from the Hospital Italiano de Buenos Aires.

Randomized patient will received a bottle of 35 pills with 1g ERN/20mg LRPT or placebo. At week 4 (± 2 days), after randomization the patient will be assessed in the outpatient clinic. Patients with good tolerance to the study medication will receive four bottles of 35 pills with 1g ERN/20mg LRPT or placebo. At week 12 (± 2 days), patients will be assessed in the outpatient clinic patients and will be crossed over to placebo or active medication. Patients will receive a bottle of 35 pills with 1g ERN/20mg LRPT or placebo. At week 16 (± 2 days), patients with good tolerance to the study medication will receive four bottles of 35 pills with 1g ERN/20mg LRPT or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Men between 21 and 75 years old.
* Very high risk patients (according NCEP-ATP III definition) with coronary heart disease (CHD) or peripheral arterial disease (PAD), documented by an angiographic study.
* Clinical stability.
* Low HDL-C plasma levels: < 40 mg/dL in men or <50 mg/dL in women in the screening and lead-in blood sample tests.
* LDL-C plasma levels between 70-100 mg/dL or non-HDL-C between 100-130 mg/dL if TG were > 200 mg/dL in the screening and lead-in blood sample tests.
* Statin based-treatment with or without ezetimibe in a stable dose in last 8 weeks.
* Women must be postmenopausal for at least 2 years and ≤ 75 years old.

Exclusion Criteria:

* Coronary event o arterial revascularization in the past 6 months.
* Uncontrolled diabetes mellitus (HbA1C > 8%).
* Acute crisis, history of gout or uric acid > 9 mg/dL.
* Thyroid stimulating hormone (TSH) outside the central laboratory's normal reference range.
* Renal insufficiency (creatinine > 1.5 mg/dL).
* Baseline alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) levels > 1.5 UNL.
* Baseline creatine kinase (CK) > 2 UNL.
* Triglycerides plasma level ≥ 500 mg/dL.
* Active fibrate therapy.
* Age > 75 years old.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Nominal change from baseline in low density lipoprotein- cholesterol (LDL-C) at 12 weeks of treatment with the extended release niacin /laropiprant combination added to usual therapy. | Week -1, baseline (week 0), week (12 ± 2 days) and week 24 (± 2days).
  Will be calculated by the Friedewald equation. With plasma triglycerides levels >400 mg/dL, LDL-C will be measured by an homogeneous method.

SECONDARY OUTCOMES:
Efficacy on other lipid variables: high density lipoprotein-cholesterol (HDL-C), triglycerides, total cholesterol (TC), TC/HDL-C ratio, apolipoprotein B (ApoB), apolipoprotein A1 (ApoA), ApoB/ApoA ratio and lipoprotein (a) [Lp(a)]. | Baseline (week 0), week 12 (± 2 days) and week (24 ± 2 days).
  TC: enzymatic method. HDL-C: homogeneous direct method. Lp(a),ApoA and ApoB: nephelometric method, using an Immage immunochemistry system (Beckman Coulter).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina